CLINICAL TRIAL: NCT07166536
Title: Characterization of Headache and Dizziness Exacerbation Following Mental Imagery in Patients With Persistent Post-Concussive Symptoms
Brief Title: Symptom Exacerbation Following Mental Imagery in Patients With Persistent Post-Concussive Symptoms
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Reuth Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0003-25-RRH
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Mild Traumatic Brain Injury, Concussion; Post Concussive Syndrome, Chronic; Post Traumatic Headache
Keywords: mild traumatic brain injury; Persistent Post-Concussion Symptoms; mental imagery; concussion
MeSH Terms: conditions — Brain Concussion; Post-Concussion Syndrome; Post-Traumatic Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mental Imagery Provocation Testing (Experimental): Provocation Test for Symptoms Using Mental Imagery:
  1. Baseline symptom intensity (dizziness/headache) will be measured using the VAS scale.
  2. Instruction to perform the movement that is hypothesized to provoke the symptom in reality for approximately 10-20 seconds
  3. Measurement of symptom intensity using the VAS scale following the provoked movement.
  4. Rest period of several minutes.
  5. Measurement of symptom intensity following rest using the VAS scale.
  6. Instruction to mentally imagine the movement or scenario hypothesized to provoke the symptom in reality for approximately 10-20 seconds
  7. Measurement of symptom intensity using the VAS scale following mental imagery.
  8. Measurement of imagery vividness using the VAS-V scale.
  Interventions: Other: Provocation Test for Symptoms Using Mental Imagery

INTERVENTIONS:
Other: Provocation Test for Symptoms Using Mental Imagery — • The mental imagery task will be guided by the examiner through continuous verbal instruction (the examiner will provide ongoing instructions throughout the entire task, not just at the beginning). During the instruction, the examiner will direct the participant's attention to visual, auditory, and proprioceptive aspects of the imagined movement or scenario. Example: "Close your eyes, and without moving your head or body at all, try to imagine that you are moving your head from side to side quickly and easily, while noticing the sensation of motion, seeing the rotation through your eyes, and feeling the acceleration of your head as it moves from side to side..."

SUMMARY:
Background: Mild Traumatic Brain Injury (mTBI) often results in persistent emotional, cognitive, and somatic symptoms-such as headaches and dizziness. These symptoms impose a significant burden, yet their underlying mechanisms remain unclear.

Predictive processing theories suggest that persistent symptoms may result from learned perceptual errors, particularly in individuals with high negative affectivity. This framework may help explain ongoing persistent post-concussive symptoms (PPCS) in the absence of identifiable pathology, which have been linked to various psychological factors.

Mental imagery (MI) is thought to engage similar predictive processes. There is evidence that MI of symptom-triggering movements may exacerbate symptoms in individuals with chronic somatic conditions. However, this phenomenon has not been studied in PPCS patients. Investigating symptom provocation through MI may yield novel insights into the neuropsychological mechanisms sustaining PPCS and potentially contribute to the development of therapeutic tools for this population.

Objectives:

1. Documenting the exacerbation of headache and dizziness following provocative mental imagery (imagery of movements or scenarios that elicit these symptoms in real life) in patients with PPCS.
2. Comparing changes in headache and dizziness after provocative MI versus neutral MI (imagery of movements or scenarios that do not elicit these symptoms in real life).
3. Comparing patients who experience symptom exacerbation following mental imagery to those who do not.
4. Describing associations between symptom exacerbation and negative affectivity, anxiety, depression, catastrophizing, and lower daily functioning.

Methods: A cross-sectional study will be conducted on adult patients experiencing PPCS following mTBI. Participants will be recruited through convenience sampling from a computerized hospital database of Reuth Rehabilitation Hospital, based on inclusion and exclusion criteria.

After signing an informed consent form, participants will be invited to attend 2 to 3 sessions, each lasting 1 to 2 hours. During these sessions, a licensed physiotherapist will conduct a comprehensive clinical assessment, including: Completion of self-report questionnaires; A vestibular examination; Anamnestic interview and clinical assessment of individual movement- and scenario-related triggers for dizziness and headaches; Symptom provocation testing using mental imagery of the identified triggers.

DETAILED DESCRIPTION:
Study Procedure

Phase 1 - Recruitment A sample will be drawn from the hospital's computerized database based on the inclusion and exclusion criteria.

Phase 2 - Patient Enrollment Potential patients will be contacted by phone and given an extensive overview of the study. They will be invited to participate in the study, and will have to arive to Reuth Rehabilitation Hospital in Tel Aviv in order to sign an informed cosent form in front of a physician that will give them an additional explanation about the study and will answer all their questions and conserns. Current patients of Reut Rehabilitation Hospital will be invited to attend research sessions during their regular treatment days. Patients who have been discharged from the hospital will be invited to participate in research sessions at their convenience, with the option to schedule the first session shortly after signing the informed consent form.

Phase 3 - Medical Record Data Collection Data extraction from patients' medical records, including demographic information, injury date and mechanism, physical and cognitive consequences, additional symptoms, imaging findings, medical history, medication use, previous treatments, and social, psychological, or psychiatric status.

Phase 4 - Clinical Assessments Assessment Session 1

* Cognitive screening test: In accordance with the Institutional Review Board (IRB) requirement, the Mini-Mental State Examination (MMSE) will be administered to provide a gross screening of cognitive status and to confirm eligibility for informed consent and study participation. Participants scoring <20 points will be excluded.
* Completion of self-reported questionnaires, including demographic information, symptoms and triggers, concussion symptomatology, dizziness-related disability, headache impact, catastrophizing, PTSD levels, anxiety, depression, negative affectivity and somatization.
* Vestibular and oculomotor assessment, including the Video Head-Impulse Test (vHIT) to rule out central and peripheral vestibular pathology, conducted by a certified vestibular physiotherapist.

Assessment Session 2

* Completion of the vestibular assessment and questionnaires (if not completed in Session 1).
* Symptom provocation test using mental imagery in a randomized order:

  * Movement mental imagery: Randomized sequence of 2 provocative movements and 2 neutral movements for each symptom (headache and/or dizziness).
  * Scenario mental imagery: Randomized sequence of 2 provocative scenarios and 2 neutral scenarios for each symptom (headache and/or dizziness).

Assessment Session 3

• Completion of pending assessments.

Phase 5 - Study Completion

ELIGIBILITY:
Inclusion Criteria:

1. Current patients of Reut Rehabilitation Hospital or individuals who were discharged from the hospital within the past 12 months.
2. Diagnosis of mild Traumatic Brain Injury, concussion, blast injury, or cervical whiplash injury.
3. More than 3 months since the event.
4. Presence of headaches and/or dizziness that began after the injury and have persisted continuously or intermittently.
5. Exclusion of other potential causes of headaches, such as non-healed fractures, chronic inflammation/infection, increased intracranial pressure, or meningeal injury.
6. Headache intensity of at least 3/10 on the VAS scale.

Exclusion Criteria:

1. Significant cognitive impairment preventing informed consent (Mini-Mental State Examination score <20 or Montreal Cognitive Assessment score <20, as per IRB requirements).
2. Diagnosed central neurological conditions such as multiple sclerosis, Parkinson's disease, stroke, or brain tumor.
3. Presence of known pyramidal or extrapyramidal neurological signs.
4. Significant language impairment interfering with communication.
5. Psychiatric disorders significantly affecting communication.
6. Use of vestibular-suppressant medication (e.g., Cinnarizine) with an inability or unwillingness to discontinue treatment 24 hours prior to testing.

Withdrawal Criteria:

1. Oculomotor dysfunction affecting multiple oculomotor functions.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-07 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Headache intensity Change | Immediately before and after the intervention at assessment session 2
  Measured on Visual Analog Scale
Dizziness intensity change | Immediately before and after the intervention at assessment session 2
  Measured on Visual Analog Scale

SECONDARY OUTCOMES:
Headache Impact on Daily life | Within 1-2 weeks before the intervention
  Headache Impact Test-6 (HIT-6): A brief assessment tool used to measure the impact of headaches on daily life. The questionnaire includes six questions addressing the frequency of functional impairment, pain intensity, and quality of life related to headaches
Post-Concussion Symptoms | Within 1-2 weeks before the intervention
  Rivermead Post-Concussion Symptoms Questionnaire (RPQ): A questionnaire assessing the severity of post-concussion symptoms. It includes 16 items where participants rate their symptoms compared to their pre-injury state on a Likert scale from 0 ("not experienced at all") to 4 ("severe problem").
Perceived disability due to dizziness | Within 1-2 weeks before the intervention
  Dizziness Handicap Inventory (DHI): A questionnaire assessing the level of disability caused by dizziness. It consists of 25 items and provides a score in percentages, where 100% indicates a high level of perceived self-disability.
Pain Catastrophizing | Within 1-2 weeks before the intervention
  Pain Catastrophizing Scale - A questionnaire assessing catastrophic thoughts related to pain, consisting of 13 items rated on a scale from 0 ("Never") to 4 ("Very much"). A high score indicates a tendency toward catastrophizing-exaggerated negative thoughts, helplessness, and magnification in response to pain.
Anxiety | Within 1-2 weeks before the intervention
  Hospital Anxiety and Depression Scale (HADS): A 14-item questionnaire assessing anxiety (HADS-A) and depression (HADS-D) in medical patients. Each subscale consists of 7 items rated on a 0-3 Likert scale, with total scores ranging from 0 to 21, where higher scores indicate greater symptom severity.
Depression | Within 1-2 weeks before the intervention
  Hospital Anxiety and Depression Scale (HADS): A 14-item questionnaire assessing anxiety (HADS-A) and depression (HADS-D) in medical patients. Each subscale consists of 7 items rated on a 0-3 Likert scale, with total scores ranging from 0 to 21, where higher scores indicate greater symptom severity.
Positive and Negative Affect | Within 1-2 weeks before the intervention
  Positive and Negative Affect Schedule (PANAS): A questionnaire assessing positive and negative emotions, consisting of 20 items divided into two subscales: positive affect and negative affect. Participants rate the intensity of emotions they experienced over a specified period on a Likert scale from 1 ("Not at all") to 5 ("Very much").
PTSD symptom levels | Within 1-2 weeks before the intervention
  Post-Traumatic Stress Disorder Checklist for DSM-5 (PCL-5): A questionnaire assessing PTSD symptoms, including 20 items where participants rate symptom severity on a Likert scale from 0 ("Not at all") to 4 ("Very much").
Somatization | Within 1-2 weeks before the intervention
  Somatization subscale of the Symptom Checklist-90-Revised (SCL-90-R): A questionnaire that assesses the presence and severity of somatic symptoms. It includes 12 items related to physical complaints such as pain, gastrointestinal issues, and cardiopulmonary symptoms. Each item is rated on a 0-4 Likert scale, with higher scores indicating greater levels of somatization.

CONTACTS AND LOCATIONS:
Overall Officials: Keren Sivan-Speier, MD, Principal Investigator — Reuth Rehabilitation Hospital
Locations (1):
- Reuth Rehabilitation Hospital, Tel Aviv, Israel

REFERENCES:
- [Background] Polinder S, Cnossen MC, Real RGL, Covic A, Gorbunova A, Voormolen DC, Master CL, Haagsma JA, Diaz-Arrastia R, von Steinbuechel N. A Multidimensional Approach to Post-concussion Symptoms in Mild Traumatic Brain Injury. Front Neurol. 2018 Dec 19;9:1113. doi: 10.3389/fneur.2018.01113. eCollection 2018. PMID 30619066
- [Background] de Neeling M, Liessens D, Depreitere B. Relationship between psychosocial and psychiatric risk factors and poor long-term outcome following mild traumatic brain injury: A systematic review. Eur J Neurol. 2023 May;30(5):1540-1550. doi: 10.1111/ene.15713. Epub 2023 Feb 15. PMID 36708085
- [Background] Dijkstra N, Bosch SE, van Gerven MAJ. Shared Neural Mechanisms of Visual Perception and Imagery. Trends Cogn Sci. 2019 May;23(5):423-434. doi: 10.1016/j.tics.2019.02.004. Epub 2019 Mar 12. PMID 30876729
- [Background] Van den Bergh O, Witthoft M, Petersen S, Brown RJ. Symptoms and the body: Taking the inferential leap. Neurosci Biobehav Rev. 2017 Mar;74(Pt A):185-203. doi: 10.1016/j.neubiorev.2017.01.015. Epub 2017 Jan 17. PMID 28108416
- [Background] Moseley GL, Zalucki N, Birklein F, Marinus J, van Hilten JJ, Luomajoki H. Thinking about movement hurts: the effect of motor imagery on pain and swelling in people with chronic arm pain. Arthritis Rheum. 2008 May 15;59(5):623-31. doi: 10.1002/art.23580. PMID 18438892